CLINICAL TRIAL: NCT03614988
Title: Comparative Evaluation of Evening Versus Morning Levothyroxine Administration in Treatment of Hypothyroidism in Elderly
Brief Title: Evaluation of Evening Versus Morning Levothyroxine Intake in Elderly
Acronym: MONIALE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 180209
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Aging; Primary Hypothyroidism; Interaction Drug Food
Keywords: Polypharmacy; Elderly
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Levothyroxine Intake First (Active Comparator): Randomized patients to receive levothyroxine in the morning and after crossover to Evening Levothyroxine Administration.
  Interventions: Other: Evening Levothyroxine Administration
- Evening Levothyroxine Intake First (Experimental): Randomized patients to receive levothyroxine in the morning and after crossover to Morning Levothyroxine Administration.
  Interventions: Other: Morning Levothyroxine Administration

INTERVENTIONS:
Other: Evening Levothyroxine Administration — Bedtime levothyroxine intake, with 60-minute meal-free interval
  Other Names: Bedtime Levothyroxine Administration
  Arms: Morning Levothyroxine Intake First
Other: Morning Levothyroxine Administration — Morning levothyroxine intake, 60 minutes before breakfast.
  Other Names: Before Breakfast Levothyroxine Administration
  Arms: Evening Levothyroxine Intake First

SUMMARY:
A study designed to compare evening versus morning levothyroxine intake in the elderly.

DETAILED DESCRIPTION:
This is a randomized crossover trial of two dosing strategies for pharmacological treatment of hypothyroidism in a sample of individuals aged 60 years or older, performed at an outpatient healthcare in a tertiary center.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years or older who consult at the Geriatrics, Endocrinology and Internal Medicine Clinic at Hospital Clinicas de Porto Alegre
* Patients diagnosed with Primary Hypothyroidism
* Patients on levothyroxine for at least 6 months
* Patients with the same dose of levothyroxine for at least 3 months

Exclusion Criteria:

* Severe Dementia
* Severe Congestive Heart Failure (NYHA IV or / and three or more hospitalizations for heart failure within 1-year interval)
* Diagnosis of Advanced Stage Neoplasia
* Diagnosis of Thyroid Cancer

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Variation in TSH (Thyroid-Stimulating Hormone) levels. | 24 weeks.
  Variation in TSH (Thyroid-Stimulating Hormone) levels after 24 weeks of levothyroxine use in the evening compared to the morning period.

SECONDARY OUTCOMES:
Prevalence of drugs with potential drug interaction with levothyroxine. | 24 weeks
  To identify the major medications that interfere with the absorption of levothyroxine.
Level of TSH (Thyroid-Stimulating Hormone) control in each group. | 24 weeks
  To compare the TSH (Thyroid-Stimulating Hormone) control efficacy between the two treatment strategies in this subgroup of participants.
TSH (Thyroid-Stimulating Hormone) levels of the patients at baseline | Baseline (0 weeks)
  To assess the TSH (Thyroid-Stimulating Hormone) levels in this sample of patients at the time of study inclusion, in order to evaluate their real life in terms of adherence and relation with polypharmacy.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Gorga Bandeira de Mello, Principal Investigator — Professor of the Post Graduate Program in Endocrinology at the Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giassi K, Piccoli V, da Costa Rodrigues T, Gorga Bandeira de Mello R. Evaluation of evening versus morning levothyroxine intake in elderly (MONIALE). Trials. 2019 Dec 17;20(1):742. doi: 10.1186/s13063-019-3816-3. PMID 31847914